CLINICAL TRIAL: NCT03176095
Title: Celiac Disease Prevention With Probiotics
Acronym: CiPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2011/335
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Celiac Disease in Children
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Active Comparator): The participants in the Probiotic group were provided with dietary supplements in the form as sachets with freeze dried bacteria (active lactobacilli culture) mixed with maltodextrin for daily intake (1 per day). The powder was dissolved in water or other non-alcoholic cold drink mixed with fruit before ingestion.
  The probiotic product consisted of two different bacterial strains.
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): The participants in the Placebo group were provided with dietary supplements in the form as sachets with maltodextrin for daily intake (1 per day).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic
  Arms: Probiotic Group
Dietary Supplement: Placebo
  Arms: Placebo Group

SUMMARY:
Background/Aim: Celiac disease is a common immune-mediated disorder, and the only currently available treatment is a gluten-free diet. Recent studies have shown several probiotics to carry properties that might positively influence the immunological activity in celiac patients.

The aim of the present study is to investigate how daily consumption of probiotics would affect levels of tissue transglutaminase autoantibodies (tTGA), markers of celiac disease autoimmunity in the periphery, as compared to placebo in children at genetic risk for celiac disease.

Methods: Between 2012 and 2015, 90 children were recruited from two ongoing prospective celiac disease screening studies at the Skåne University Hospital, Sweden. Participants were randomized to either daily consumption of 2 lactobacilli strains or placebo for the duration of 6 months.

Blood samples were drawn at 0, 3 and 6 months and analyzed for both IgA-tTGA and IgG-tTGA using radioligand binding assays.

ELIGIBILITY:
Inclusion Criteria:

* Carrier of any of the HLA-types DQ2 and/or DQ8 associated with celiac disease.
* Screened positive for tissue transglutaminase autoantibodies (tTGA) in at least 2 consecutive blood draws (<30U/ml).
* No celiac disease diagnose
* Currently on a normal gluten-containing diet

Exclusion Criteria:

* Screened positive for Type 1 diabetes associated autoantibodies (GADA, IAA, IA-2A, ZnT8A).

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2015-08-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Tissue transglutaminase autoantibodies (tTGA) | 6 months
  To study levels of tTGA in children with ongoing celiac disease autoimmunity

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Agardh, MD, PhD, Principal Investigator — Lund University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Auricchio R, Troncone R. Can Celiac Disease Be Prevented? Front Immunol. 2021 May 14;12:672148. doi: 10.3389/fimmu.2021.672148. eCollection 2021. PMID 34054850
- [Background] Jedwab CF, Roston BCMB, Toge ABFS, Echeverria IF, Tavares GOG, Alvares MA, Rullo VEV, Oliveira MRM. The role of probiotics in the immune response and intestinal microbiota of children with celiac disease: a systematic review. Rev Paul Pediatr. 2021 Sep 1;40:e2020447. doi: 10.1590/1984-0462/2022/40/2020447. eCollection 2021. PMID 34495279
- [Result] Hakansson A, Andren Aronsson C, Brundin C, Oscarsson E, Molin G, Agardh D. Effects of Lactobacillus plantarum and Lactobacillus paracasei on the Peripheral Immune Response in Children with Celiac Disease Autoimmunity: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Nutrients. 2019 Aug 16;11(8):1925. doi: 10.3390/nu11081925. PMID 31426299
- [Result] Oscarsson E, Hakansson A, Andren Aronsson C, Molin G, Agardh D. Effects of Probiotic Bacteria Lactobacillaceae on the Gut Microbiota in Children With Celiac Disease Autoimmunity: A Placebo-Controlled and Randomized Clinical Trial. Front Nutr. 2021 Jun 25;8:680771. doi: 10.3389/fnut.2021.680771. eCollection 2021. PMID 34249990
- [Derived] Jenickova E, Andren Aronsson C, Mascellani Bergo A, Cinek O, Havlik J, Agardh D. Effects of Lactiplantibacillus plantarum and Lacticaseibacillus paracasei supplementation on the faecal metabolome in children with coeliac disease autoimmunity: a randomised, double-blinded placebo-controlled clinical trial. Front Nutr. 2023 Jul 6;10:1183963. doi: 10.3389/fnut.2023.1183963. eCollection 2023. PMID 37485388